CLINICAL TRIAL: NCT02815566
Title: Bone Health in Aging HIV Infected Women: Improvement or Prevention of Changes in Bone Mineral Density by Switching Antiretroviral Agents. Is There an Optimal Time to Intervene?
Brief Title: Bone Health in Aging HIV Infected Women
Acronym: BEING
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: University of Modena and Reggio Emilia (Other); San Raffaele University Hospital, Italy (Other); Gilead Sciences (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, University Health Network-Toronto General Hospital, Professor of Medicine, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 16-5543; IN-CA-311-3963 (Other Grant/Funding Number: Gilead)
Record Dates: First submitted 2016-06-22; First posted 2016-06-28 (Estimated); Results first posted 2023-01-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Osteoporosis; HIV; Menopause
Keywords: kidney, antiretroviral agent, tenofovir, osteoporosis, women
MeSH Terms: conditions — Osteoporosis | interventions — emtricitabine tenofovir alafenamide; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Immediate switch (Experimental): Open label tenofovir-alafenamide (25/10mg)-emtricitabine (200mg) tablet once daily by mouth for 96 weeks
  Interventions: Drug: tenofovir-alafenamide-emtricitabine
- delayed switch (Active Comparator): Open-label tenofovir (300mg)-emtricitabine (200mg) tablet once daily by mouth for 48 weeks followed by open label tenofovir-alafenamide (25/10mg)-emtricitabine (200mg) tablet once daily by mouth for an additional 48 weeks
  Interventions: Drug: tenofovir-emtricitabine

INTERVENTIONS:
Drug: tenofovir-alafenamide-emtricitabine — comparison of tenofovir-emtricitabine and tenofovir-alafenamide-emtricitabine on bone mineral density
  Other Names: Descovy
  Arms: Immediate switch
Drug: tenofovir-emtricitabine — comparison of tenofovir-emtricitabine and tenofovir-alafenamide-emtricitabine on bone mineral density
  Other Names: Truvada
  Arms: delayed switch

SUMMARY:
Design: Open-label randomised multicenter international strategic trial of older women on combination antiretroviral therapy (cART) containing tenofovir-emtricitabine (TDF/FTC) with HIV RNA suppression for > 6 months to : 1. Immediate switch of TDF/FTC to tenofovir alafenamide-emtricitabine (TAF/FTC) while continuing the third antiretroviral agent.; 2. Delayed switch; with switch of TDF/FTC to TAF/FTC at 48 weeks while continuing the third agent. Follow up of all subjects to 96 weeks.

Subject Population: The anticipated sample size is 128 HIV infected women aged 45-55 years (peri or early post menopause). .

Primary endpoint: Percentage change from baseline bone mineral density (BMD) at the lumbar spine at weeks 48 and 96.

Secondary Endpoints: BMD change at hip, trabecular bone score, estimated bone strength by high resolution peripheral quantitative computerized tomography (HR-pQCT), muscle quality, geriatric assessment; biomarkers of bone, immune activation and inflammation; HIV viral suppression; safety, lipid and renal function, cardiovascular risk scores at weeks 48 and 96.

Expected Outcomes: To determine if a switch from TDF/FTC to TAF?FTC improves BMD to a degree correlating with a decreased risk of fragility fracture in aging HIV infected women. Secondary outcomes will assess bone strength using new imaging modalities, timing of switch, and renal health. This data will be used by health policy makers and providers to determine the proper use of TAF/FTC in the aging HIV population.

DETAILED DESCRIPTION:
A Randomized controlled clinical trial (RCT) of immediate vs delayed switch from TDF/FTC to TAF/FTC to define the impact of switching ARV on BMD in different stages of the aging trajectory in HIV infected women. Included is a geriatric assessment based on the conceptualization of health transition across menopause.

Study Hypothesis: The primary hypothesis is that switching from TDF/FTC will improve BMD to a degree that correlates with a lower fracture risk in aging HIV+ women. We will further explore our theory that the impact is greater in those in the early stages of menopause and in those who also receive a protease inhibitor (PI) as the third antiretroviral agent (ARV).

Primary objectives: To determine if: 1. Switching HIV+ women on TDF/FTC to TAF/FTC increases BMD at the spine at 48 weeks relative to those who continue TDF/FTC 2. To determine if any observed improvements continue or stabilize in the year after switch.

Hypothesis generating objectives: To determine if the effect of switching from TDF/FTC to TAF/FTC on BMD varies by stage of menopause and by third ARV.

Study design: This study is double blind placebo controlled randomised, 1:1, multicentre strategic trial. Patients will be randomised to immediate vs delayed switch, with randomization allocation arranged to minimize differences between treatment group with respect to stage of menopause (peri- menopause vs early post menopause) and site. Study population: HIV positive women who are in the peri-menopausal period or those within 10 years post menopause to capture those with greatest risk of BMD loss. As menopause typically occurs earlier in HIV + women we include those aged 45-55 years. They must be on a cART regimen containing TDF/FTC with HIV RNA <50 c/ml for at least 6 months.

Intervention:

1. Immediate switch of TDF/FTC to TAF/FTC while maintaining the third ARV agent.
2. Delayed switch of TDF/FTC to TAF/FTC at 48 weeks while maintaining the third ARV agent.

Randomization: A computer-generated randomization list will be prepared prior to study onset by a statistician unassociated with the study. Randomization will be stratified by study centre.

Primary endpoint: Comparison of the immediate vs delayed group in the % change from baseline in BMD at the lumbar spine at week 48 and 96.

Secondary endpoints: Will compare changes between the immediate and delayed group from data collected at screening or baseline and weeks 48 and 96.

* change from baseline in BMD at hip Changes in Bone architecture as determined by Trabecular bone scan (TBS) and HRpQCT (high resolution peripheral quantitative computerized tomography) (Toronto site) Changes in 10 year fracture risk determined by country specific FRAX® (fracture risk assessment) calculator
* with HIV-1 RNA <50 c/ml Change from baseline in geriatric functional measures: frailty, performance and balance Change from baseline in muscle quality: Sarcopenia - grip strength measured by a Dynamometer Change from baseline in lipid values and Framingham cardiovascular risk scores Changes in renal tubular and glomerular function: GFR (glomerular filtration rate), Creatinine, urine albumin /creatinine and protein/creatinine, glucosuria Safety (clinical and laboratory adverse events) Changes in biomarkers of inflammation, coagulation and bone metabolism Tolerability (EuroQoL questionnaire)

ELIGIBILITY:
Inclusion Criteria:

1. Biological female aged 40-60
2. Documented HIV-1 infection
3. Peri-menopausal ( as documented by history).
4. Signed Informed Consent Form and willing to comply with the protocol.
5. Receiving a cART regimen containing a ritonavir boosted PI (darunavir, atazanavir, lopinavir,) or an NNRTI (efavirenz, nevirapine or rilpivirine) or an integrase inhibitor (dolutegravir or raltegravir or elvitegravir) in combination with TDF-FTC for > 24 weeks.
6. Stable viral suppression (plasma HIV-RNA<50 copies/mL for > 24 weeks). Single viral blip <500/ml allowed if re-suppresses.
7. If of childbearing potential, is using effective birth control methods and is willing to continue during the trial.
8. Women will be assessed for vitamin D and calcium dietary intake; if inadequate for age, supplements will be recommended.

Exclusion Criteria:

1. HIV-2
2. High 10-year fracture risk at baseline ( > 20%) based on country specific FRAX
3. Current treatment with active bone medications- bisphosphonates, denosumab, calcitonin, raloxifene, teriparatide, strontium
4. Current use of systemic steroids ( inhaled steroids permitted) or chemotherapeutic agents
5. Acute viral hepatitis
6. Chronic hepatitis C with liver transaminases >5 x ULN or expected to require treatment for hepatitis C during the trial period.
7. Any investigational ARV within 30 days.
8. Dialysis or renal insufficiency (creatinine clearance < 50ml/min)
9. History of decompensated liver disease (AST or ALT≥5x the upper limit of normal (ULN) or ALT ≥ 3 x ULN and bilirubin ≥ 1.5 x ULN with > 35% direct bilirubin), or the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices.
10. Pregnant or breastfeeding
11. Screening blood result with any grade 3/4 toxicity according to Division of AIDS (DAIDS) grading scale, except: asymptomatic grade 3 amylase, creatinine phosphokinase, or lipid elevation.
12. Any condition (including illicit drug use or alcohol abuse) or lab results which, in the investigator's opinion, interfere with assessments or completion of the trial.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-12 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: sharon walmsley, MD, Principal Investigator — University Health Network, Toronto
Locations (7):
- Canada (5):
  - Vancouver ID Research and Care Centre, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
- Italy (2):
  - Ospedale San Raffaele, Milan
  - Università degli Studi di Modena e Reggio Emilia, Modena

IPD SHARING:
Plan to Share IPD: Yes
Information on viral load, toxicity and bone scans will be available to treating physicians

REFERENCES:
- [Result] Walmsley S, Clarke R, Lee T, Singer J, Cheung AM, Smaill F, De Pokomandy A, Trottier S, Messina E, Guaraldi G. BEING: Bone Health in Aging Women with HIV: Impact of Switching Antiretroviral Therapy on Bone Mineral Density During the Perimenopausal Period. AIDS Res Hum Retroviruses. 2023 Apr;39(4):204-210. doi: 10.1089/AID.2022.0106. Epub 2023 Jan 20. PMID 36511389

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Immediate Switch | Delayed Switch
Started | 19 | 15
Completed | 17 | 13
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Switch | Delayed Switch | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.0 (3.1) | 48.8 (2.9) | 50.6 (3.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 10 | 20
  White | 8 | 5 | 13
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 13 | 11 | 24
  Italy | 6 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Bone Mineral Density From Baseline at the Lumbar Spine
Description: The outcome measures presented are descriptive as enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results. There are limited results at the week 48 timepoint due to the COVID pandemic.
Time Frame: Baseline, 48 weeks and 96 weeks
Population: Thirty-four women enrolled: 19 in the immediate and 15 in the delayed switch arm between Sept 2017 and April 2019; 30 completed the 96-week protocol. The study closed to follow up March 2021. Two participants in the delayed arm inadvertently switched to TAF at baseline and one participant in the delayed arm remained on TDF for the entire 96 weeks.
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 19 | 15
Percent Change
  48 weeks: number analyzed (Participants) | 13 | 10
  48 weeks | 1.97 [-1.15 to 5.49] | -2.32 [-5.11 to 0.19]
  96 weeks: number analyzed (Participants) | 18 | 11
  96 weeks | 2.33 [0 to 4.51] | 0.7 [-3.19 to 2.47]

2. Secondary Outcome: % Change in Bone Mineral Density From Baseline at the Femoral Neck
Description: as for outcome 1
Time Frame: Baseline, 48 weeks and 96 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Percent Change
Arm/Group | Immediate Switch | Delayed Switch
Number analyzed (Participants) | 19 | 15
Percent Change
  48 weeks: number analyzed (Participants) | 13 | 10
  48 weeks | 1.46 [-2.95 to 3.18] | 0.22 [-2.83 to 3.64]
  96 weeks: number analyzed (Participants) | 18 | 11
  96 weeks | 2.33 [0 to 4.51] | 0.70 [-3.19 to 2.47]

ADVERSE EVENTS:
Time Frame: 96 Weeks
Description: Any grade 3 or 4 AE and all fractures that occurred from screening to the end of the study (Week 96 or Early Termination) was captured and recorded.
Groups:
- Delayed Switch: Open-label tenofovir (300mg)-emtricitabine (200mg) tablet once daily by mouth for 48 weeks and
  tenofovir-emtricitabine: comparison of tenofovir-emtricitabine and tenofovir-alafenamide-emtricitabine on bone mineral density
- Delayed Switch: Open label tenofovir-alafenamide (25/10mg)-emtricitabine (200mg) tablet once daily by mouth for an additional 48 weeks.
  tenofovir-emtricitabine: comparison of tenofovir-emtricitabine and tenofovir-alafenamide-emtricitabine on bone mineral density
Arm/Group | Immediate Switch | Delayed Switch | Delayed Switch
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 2/19 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Switch (N=19) | Delayed Switch (N=15) | Delayed Switch (N=15)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
HIV Encephalitis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Enrollment was a challenge and did not reach the target subject number and was insufficient to produce statistically reliable results. This was primarily due to long delays in study start-up associated with contract negotiations. During the delays, most eligible participants switched to a TAF based regimen outside of the study. The COVID pandemic prevented enrollment of additional participants. The study was closed to futility on the recommendation of the DSMB

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02815566/Prot_SAP_000.pdf